CLINICAL TRIAL: NCT05059145
Title: A RCT for Chlorhexidine Gluconate as Treatment and Prophylaxis for Recurrent Vulvovaginal Candidiasis
Brief Title: A Clinical Trial for Chlorhexidine as Treatment for Vulvovaginal Candidiasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Nina Bohm-Starke, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chlorhex-KKDS-2021
Record Dates: First submitted 2021-02-19; First posted 2021-09-28 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Candidiasis, Vulvovaginal
Keywords: Recurrent vulvovaginal candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — chlorhexidine gluconate; Fluconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine gluconate, 1% vaginal cream (Experimental): 8 ml vaginal cream every night for a week and then prophylactic treatment with 8 ml/week for another 11 weeks
  Interventions: Drug: Chlorhexidine Gluconate
- Fluconazole, 150 mg oral capsule (Active Comparator): Fluconazole150 mg (oral capsule) every 3 days for the first 3 doses, then prophylactic treatment with 150 mg/week for another 11 weeks
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Vaginal cream 1%
  Other Names: Hibitane vaginal cream
  Arms: Chlorhexidine gluconate, 1% vaginal cream
Drug: Fluconazole — 150 mg oral capsule
  Arms: Fluconazole, 150 mg oral capsule

SUMMARY:
The overall aim of this study is to investigate if vaginally applied 1% chlorhexidine gluconate (CHG) could be an alternative treatment to oral fluconazole (FLZ), both during an acute episode and as prophylaxis, against recurrent infections of vulvovaginal candidiasis (RVVC).

RVVC is very common in fertile women. Up to six months of treatment with FLZ is recommended for RVVC. Over the last ten years, the use of FLZ has increased markedly in many countries. No major problems have been noted with resistance development, but there is concern that this will occur in the future and alternative treatments are requested. In recent years, it has emerged that flukonazol interacts with several different types of drugs that are common in the patient group; several antidepressants, pain relief at dysmenorrhea (NSAID) and oral contraceptives to name a few.

In Sweden an over-the-counter vaginal cream consisting of 1% chlorhexidine gluconate (Hibitane®) is available with the indication antiseptic use in vaginal examinations, especially during childbirth. The product has been used for a long time in various gynecological and obstetric surgical procedures. Hibitane® is approved during pregnancy and the cream is usually well tolerated.

The research group has previously done an in vitro study in which we analyzed the effect of FLZ and CHG's ability to kill fungal cells and to break down existing biofilm or prevent new biofilm formation. The biofilm formation is an important stage for the fungal cells to attach to surfaces such as skin and mucosa and is considered a first step in the development of an infection. In the biofilm, the fungus can hide from the immune system and also to some extent for various treatments aimed against the fungus. The results of the study showed that CHG was better than FLZ both at killing the fungal cells and preventing new biofilm from forming and dissolving already established "old" biofilm. This effect is absolutely crucial for successful treatment with antimycotics. These encouraging results form the basis of the planned study.

If CHG is at least as effective as FLZ with little impact on vaginal lactobacillus, with high tolerability and without cytotoxic effect on epithelial cells, the results of the study might lead to major benefits to the patients with reduced risk of systemic side effects such as drug interactions, development of drug resistance and reduced drug costs.

DETAILED DESCRIPTION:
The study is a 6 months clinical Phase II trial to compare if 1% chlorhexidine gluconate vaginal cream (Hibitane®) is at least as effective and safe as fluconazole (reference treatment) for culture-verified recurrent vulvovaginal candidiasis. The study is a randomized open non-inferiority trial with parallel treatment groups. The trial is not possible to blind for neither participants nor investigators due to the differences between study treatments. There is low risk of bias since the primary outcome variable is objective (negative vaginal culture for Candida albicans).

The participants will be randomization to;

* Investigational medication with Hibitane® vaginal cream 8 ml every night for a week and then prophylactic treatment with 8 ml/week for another 11 weeks or
* Reference treatment with Fluconazole® 150 mg (oral capsule) every 3 days for the first 3 doses, then prophylactic treatment with 150 mg/week for another 11 weeks.

The randomization ratio between the treatment groups will be 1:1. A computer generated block randomization of 15 participants will be performed by the research midwife. Allocation to the study medications will be carried out via opening of opaque sealed envelopes in consecutive order. All women will be identified through a patient log with name and Swedish personal identification number and the randomization number. The randomization number will be used on all paper and CRFs.

Five research visits are planned:

Visit 1 Screening - oral and written study information, signing of informed consent, vaginal culture for Candida albicans and chlamydia/gonorrhea (PCR test).

Visit 2 Inclusion (baseline), within 1 week after Visit 1. Control for inclusion/exclusion criteria, randomization to study medication after positive culture for Candida albicans and negative chlamydia/gonorrhea (PCR test) - health survey, control of concomitant medications, examination, pregnancy test and control of adequate contraceptive methods to avoid pregnancy throughout the study.

Visit 3 1 week (+2 days) after completed treatment. Control of AE, culture for Candida albicans and examination.

Visit 4 After 12 weeks (+ 1 week) from inclusion when prophylactic treatment is completed. Control of AE and relapses, culture for Candida albicans and examination.

Visit 5 Follow-up 6 months (+ 1-2 weeks) from baseline/inclusion. Control of AE and relapses, culture for Candida albicans and examination. End of study.

A weekly web-based dairy (eCRF (Entermedic)) will be used for follow-up of treatment compliance, efficacy and adverse events. During the prophylactic treatment (Visits 2-3) and during the observational phase of the study (Visit 4-5), the participants are asked to report any suspicious relapses in the dairy and contact the research midwife if needed. They will also receive equipment for vaginal cultures that can be used for self-sampling at home to detect true relapses. In case of positive cultures for Candida albicans, they will be offered the same medication as previously used in the study if the treatment was effective and no adverse events occurred. Otherwise, an individual treatment option will be used.

The end of study is defined as completion of the last visit of the last subject. The sponsor and the investigators reserve the rights to discontinue the study at any time for safety reasons or other reasons jeopardizing the justifications of the study.

Supply, labelling, handling and storage:

Chlorhexidine gluconate (Hibitane®) vaginal cream is commercially available in Sweden and will be prescribed from the hospital pharmacy for each participant. It will be stored and kept according to the instructions of the manufacturer.

* Participants randomized to Hibitane® will receive a bottle (250ml) with the vaginal cream together with 10 ml syringes for vaginal administration. The Hibitane® bottle can be stored in the fridge at home between use. Women will receive specific written information as well as oral information on how to self-administer drug vaginally with the syringe.
* Participants randomized to Fluconazole® will receive 14 oral capsules of 150 mg according to the dosage describe above.

Compliance:

Compliance will be evaluated at the follow up visits and the participants will fill out a dairy how the study medications have been taken.

Data collection and data handling:

Every participant will be given an individual, study specific number (i.e. study identifying code) at the time of inclusion. A code key with each individual personal data connected to the identifying code will be created (i.e. patient identification log) and stored separately at the research department at the department of Obstetrics and Gynecology, Danderyd Hosptial, Stockholm, Sweden.

Data will be recorded on individual printed case report forms (CRFs) after which they will be entered into a computerized database before statistical analyses. The database will contain information on demographic variables, type of treatment and measurements in addition to the variables above.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* A history of > 2 candida infections the last year
* Symptoms of acute vulvovaginal candida infection
* Culture verified infection with Candida albicans
* Adequate contraceptive method
* Able to understand oral and written information in Swedish
* The subject has given written consent to participate in the study

Exclusion Criteria:

* Severe somatic or mental illness (including liver and kidney failure and cardiac disease)
* Immunosuppressive medication
* Pregnancy
* Lactation
* Other ongoing gynecological infections
* Allergy to fluconazole or chlorhexidine gluconate
* Citalopram or other medication that might have impact on the QT interval (terfenadin, cisaprid, astemizol, pimozid, kinidin, erythromycin, halofantrin, amiodaron)
* Participation or recent participation (30 days) in a clinical study with an investigational product. Previous participation in this study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women in each group that has cleared the vulvovaginal infection | Up to 10 days
  Negative vaginal culture for Candida albicans

SECONDARY OUTCOMES:
Prophylactic effect | 6 months
  Proportion of women with negativ vaginal culture for Candida albicans at follow ups
Adverse events | 6 months
  Proportion of women i each treatment arm repoting AEs
Symptom score | 6 months
  Proportion ov women with symptom score >2 of composite index 0-5 (typical discharge, itching, dryness of the skin/mucosa, burning and pain)
Examination score | 6 months
  Proportion ov women with examination score >2 of composite index 0-5 (redness skin/mucosa, typical discharge, dry skin/mucosa, fissures in skin/mucosa, visible candida hyphae in wet mount)
Vaginal lactobacillus content | 6 months
  Proportion of women with reduced vaginal lactobacilli content in vaginal smears measured by a semi-quantitative method as normal or reduced quantity.
Infection relapse | 6 months
  Proportion of women in each treatment arm with relapses of Candida albicans infection

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin Alvendal, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd Hospital, Dep. of Obstetrics and Gynecology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No